CLINICAL TRIAL: NCT07259967
Title: Laterality Success Determination of Microscopic Testicular Sperm Extraction in Non Obstructive Azoopsermia Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mohamed diab mohamed ramadan, Assistant Lecturer, Assiut University
Other Study IDs: Laterality of micro TESE
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Testicular Sperm Extraction in Azoospermic Patients
Keywords: azoospermia; TESE
MeSH Terms: conditions — Azoospermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Testicular sperm extraction — Bilateral Testicular sperm extraction done under microscopic guidance for non obstructive azoospermic patients

SUMMARY:
Determination of percentage of successful sperm retrieval in single testis in cases who will do bilateral TESE and identification factors mostly associated with successful sperm retrieval

DETAILED DESCRIPTION:
Male infertility is defined as the failure of pregnancy within 12 months despite the presence of a fertile female partner and coitus via a normal vaginal route without contraception. The microscopic absence of spermatozoa in the ejaculate in at least two semen analysis samples is defined as azoospermia. Azoospermia plays a role in the etiology of male infertility with a rate of 10-15% . Azoospermia is divided into two subgroups: obstructive azoospermia (OA) and non obstructive azoospermia (NOA). NOA is detected in 60% of patients with azoospermia. The etiopathogenesis of NOA includes genetic disorders, Y chromosome microdeletions, testicular torsion, cryptorchidism, toxins, radiation and idiopathic factors. Although many techniques including Percutaneous Sperm Aspiration , Testicular Sperm Aspiration , Conventional Testicular Sperm Extraction , Microdissection Testicular Sperm Extraction (MD-TESE) have been used to detect sperm in patients with NOA, MD-TESE is currently accepted as the method with the highest sperm retrieval rate with the least complications and tissue loss. However, no standard approach is available for searching for appropriate tubules during the MD-TESE procedure . A limited number of studies are available in the literature on whether the testicle should be explored transversely or longitudinally, bilaterally or unilaterally, to increase the sperm detection rate in MD-TESE, and there is still no standard systematic procedure for MD-TESE today to minimize the possibility of missing appropriate tubules and obtaining sperm. Furthermore, despite the presence of studies in the literature indicating that parameters such as hormonal values, testicular volume, genetics, age, environmental factors, varicocele and cryptorchidism predict the possibility of finding sperm before the MD-TESE procedure, none of these parameters have a definite predictive value on sperm finding . The present study aims to evaluate if there is difference in testicular sperm retrieval in patients with non obstructive azoospermia in TESE between right and left testes.

ELIGIBILITY:
Inclusion Criteria:

* • Male patients diagnosed as non obstructive azoospermia.

  * Will do bilateral TESE.

Exclusion Criteria:

* • Obstructive azoospermia.

  * Incomplete medical record .
  * Prior testicular Trauma.

Ages: 20 Years to 60 Years | Sex: Male
Age Groups: Adult
Study Population: Male patients diagnosed as non obstructive azoospermia and will do bilateral TESE.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
percentage of successful sperm retrieval in single testis in cases who will do bilateral TESE. | 1 day Postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Diab Mohamed Ramadan, Master, Principal Investigator — Assiut University

REFERENCES:
- [Result] Raman JD, Schlegel PN. Testicular sperm extraction with intracytoplasmic sperm injection is successful for the treatment of nonobstructive azoospermia associated with cryptorchidism. J Urol. 2003 Oct;170(4 Pt 1):1287-90. doi: 10.1097/01.ju.0000080707.75753.ec. PMID 14501743
- [Result] Levin HS. Testicular biopsy in the study of male infertility: its current usefulness, histologic techniques, and prospects for the future. Hum Pathol. 1979 Sep;10(5):569-84. doi: 10.1016/s0046-8177(79)80100-8. PMID 43278
- [Result] Witt MA, Elsner C, Kort HI, Massey JB, Mitchell-Leef D, Toledo AA, Tucker MJ. A live birth from intracytoplasmic injection of a spermatozoon retrieved from testicular parenchyma. J Urol. 1995 Sep;154(3):1136-7. No abstract available. PMID 7637066
- [Result] Ichioka K, Matsui Y, Terada N, Negoro H, Goto T, Ogawa O. Three-dimensional simulation analysis of microdissection testicular sperm extraction for patients with non-obstructive azoospermia. Andrology. 2020 Sep;8(5):1214-1221. doi: 10.1111/andr.12812. Epub 2020 May 18. PMID 32374923